CLINICAL TRIAL: NCT03664843
Title: A Prospective Multicenter Study of Longitudinal Monitoring in Treated Stage III-IV Lung Cancer Patients by Circulating Tumor DNA
Brief Title: Circulating Tumor DNA Longitudinal Monitoring in Stage III-IV Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Hospital of Shijiazhuang City (Other)
Collaborators: Peking University People's Hospital (Other); Tianjin Medical University General Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Affiliated Hospital of Hebei University (Other); Hebei Medical University Fourth Hospital (Other); Xingtai People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PTH01801
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma; Non-small Cell Lung Cancer; Lung Neoplasm
Keywords: circulating tumor DNA; lung cancer; surveillance; longitudinal monitoring; lead time
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue and blood samples were collected from each patient. Histological specimens (fresh or paraffin blocks) of all enrolled patients before treatment need to be obtained, and according to different adjuvant therapy, blood samples were collected at a series of specific scheduled time-points
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The chemotherapy cohort: Blood samples for ctDNA and biomarkers analysis are collected at before chemotherapy and at a series of scheduled time-points after chemotherapy , with serial two-weekly blood samples collected from a subset of patients. Meanwhile, imaging technology such as CT scan detection would be performed.
- The radiotherapy cohort: Blood samples for ctDNA and biomarkers analysis are collected at before radiotherapy and at a series of scheduled time-points after radiotherapy, with serial two-weekly blood samples collected from a subset of patients. Meanwhile, imaging technology such as CT scan detection would be performed.
- The targeted therapy cohort: Blood samples for ctDNA and biomarkers analysis are collected at before targeted therapy and at a series of scheduled time-points after targeted therapy, with serial two-weekly blood samples collected from a subset of patients. Meanwhile, imaging technology such as CT scan detection would be performed.

SUMMARY:
Conduct a prospective study in multicenter to confirm the value of circulating tumor DNA in longitudinal monitoring of stage III-IV lung cancer patients.

DETAILED DESCRIPTION:
The study consists of two phases, the first stage is the exploratory stage of blood collection point which is the appropriate effective time after chemotherapy, radiotherapy, targeted therapy. The second phase, which is the expansion of the first phase, is to determine the precise leading time of ctDNA relative to tumor biomarkers or image evaluation in determining the efficacy of advanced NSCLC cancer therapy. Both stages were divided into three subgroups: the chemotherapy group, the radiotherapy group, and the targeted therapy group.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years old;
2. Patients with stage III-IV NSCLC;
3. Have the tissue specimens (fresh or wax blocks) before this treatment;
4. PS<=2 in radiotherapy/ chemotherapy group; PS<=3 in targeted therapy group
5. Signing informed consent;

Exclusion Criteria:

1. Multiple primary lung cancer;
2. Incorporating any unstable systemic disease;
3. Histology is not NSCLC;
4. Unqualified blood samples;
5. Patients lacking any one of the detection points.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be drawn from Oncology Department of multicenters. The enrolled patients must be patients with stage III-IV NSCLC according to the 8th edition of the TNM Classification of the International Association for the Study of Lung Cancer (IASLC), must be greater than 18 years old and must have the tissue specimens (fresh or wax blocks) before this treatment. The exclusion criteria are as followed: (1) Multiple primary lung cancer;(2) Incorporating any unstable systemic disease; (3) Histology is not NSCLC; (4)Unqualified blood samples; (5) Patients lacking any one of the detection points. All of the patients signing informed consent were not involved in the recruitment and conduct of the study
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
ctDNA effective time | 6 months
  To explore the appropriate chemo/ radio/ target effective time (CET/RET/TET) through measurement and monitoring of ctDNA after anti-cancer therapies in advanced NSCLC.
ctDNA leading time | 1 year
  To investigate the precise leading time for ctDNA compared to conventional biomarker or image evaluation in detecting disease recurrence after radiotherapy, chemotherapy, or targeted therapy respectively.

SECONDARY OUTCOMES:
Assess the accuracy of ctDNA | 1 year
  To assess the accuracy of ctDNA when imaging undetectable or difficult to assess
Compared to conventional image | 1 year
  Compared to conventional image evaluation, to determine the consistency of ctDNA in treatment response of measurable lesion after radiotherapy, chemotherapy, or targeted therapy respectively
Compared to traditional tumor markers | 6 months
  To explore the consistency for ctDNA in determining the efficacy of advanced NSCLC compared to tumor markers after radiotherapy, chemotherapy, or targeted therapy respectively

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M.D., Principal Investigator — The First Hospital of Shijiazhuang; Jun Wang, M.D., Study Chair — Peking University People's Hospital; Kezhong Chen, M.D., Study Director — Peking University People's Hospital
Locations (8):
- China (8):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - The First Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Handan Downtown Hospital, Handan, Heibe
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided